CLINICAL TRIAL: NCT03194074
Title: Early Cognitive Function and Recovery in Elderly Patients After Laser Laryngeal Surgery: Desflurane-based vs Propofol-based Anesthesia
Brief Title: Early Cognitive Function in Elderly Patients After Laser Laryngeal Surgery: Des vs Prop
Acronym: POCDLLS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Xia Shen, Vise Director of Department of Anesthesiology, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: POCD-DesProp
Record Dates: First submitted 2017-06-17; First posted 2017-06-21 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Cognition Disorders in Old Age
Keywords: Laser Laryngeal Surgery; Desflurane; Propofol
MeSH Terms: interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- propofol group (Experimental): Propofol/remifentanil-based general anesthesia.
  Interventions: Drug: Propofol
- desflurane group (Experimental): Desflurane/remifentanil-based general anesthesia.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Propofol — In propofol/remifentanil group, propofol at a rate 75~150 µg/kg/min and remifentanil at 0.1-0.3 µg/kg/min are maintained throughout surgery.
  Other Names: Propofol injection from AstraZeneca
  Arms: propofol group
Drug: Desflurane — In desflurane/remifentanil group, desflurane at end tidal concentration at 0.7~1.0 minimum alveolar concentration (MAC) and remifentanil 0.1-0.3 ug/kg/min are used.
  Other Names: Suprane from Baxter
  Arms: desflurane group

SUMMARY:
Postoperative cognitive impairment is one of the most common complications in elderly surgical patients. Laser laryngeal surgery is a short procedure, but characterized by high risk of disastrous airway fire. So the recommended oxygen concentration is less than 30%. For elderly patients, because of preoperatively declined cardiovascular and lung function and cognitive function, there is a potential that intraoperative low oxygen concentration may lead to drop of arterial oxygen tension, decrease of brain oxygenation, and exacerbate brain function impairment. Intravenous anesthesia and inhalation anesthesia is two commonly used technique for general anesthesia. Consequently, we carry out this study to identify whether different classes of anesthetics can affect postoperative cognitive function in old patient undergoing laser laryngeal surgery.

DETAILED DESCRIPTION:
The allocation sequence is generated by computer random number generation, and the allocation is placed in sequentially numbered opaque sealed envelopes by a non-investigator. Enrolment and data collection are performed by trained research staff who are not involved in the care of the patients. The treating clinicians are not blinded to the assignment group, but all other staff involved in both the collection and collation of data, and administration of neurocognitive testing, are blinded to group allocation

The primary measurement is the MMS scores. The secondary measurements are intraoperative desaturation score (multiplying Spo2 < 90% by time (seconds)), extubation time, orientation time, and time to discharge from the post-anaesthesia care unit (PACU).

A sample size of 35 was determined by using a power analysis based on the assumptions that the incidence of postoperative cognitive impairment in adult after otorhinolaryngological surgery would be as high as 50 %, b) a 70% reduction (from 50% to 15%) would be of clinical significance, and c) α= 0.05, β= 0.2.

The continuous variables were expressed as means ± standard deviation (SD) whereas categorical variables were expressed as frequency and percentage for data description.

The outcome of interest is cognitive decline. A Generalized estimating equation (GEE) model with compound symmetry covariance structure was constructed to compare differences between two treatments with different time points as the repeated factors. As the effect of treatments may vary across different time points, an interaction between treatments and time was included in the model. Bonferroni-corrected post hoc test was conducted to adjust the observed significant level for multiple comparisons if the null hypothesis was rejected.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laser laryngeal surgery under general anesthesia with either Propofol or desflurane based technique.

Exclusion Criteria:

* Patients with cardiac, pulmonary, hepatic, or renal dysfunction, epilepsy, or uncontrolled hypertension, or those taking medications that influence the central nervous system, are excluded from the study. Patients who show obvious alteration of mental status, or refuse to participate, are also excluded from the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change of Mini-Mental State (MMS) test score | Change of MMS score between two time points (the day before surgery and 30min postoperatively
  Change of 30-point questionnaire that is used to measure cognitive impairment before and after surgery

SECONDARY OUTCOMES:
Change of Mini-Mental State (MMS) test score | Change of MMS score between two time points (the day before surgery and 1h postoperatively
  Change of 30-point questionnaire that is used to measure cognitive impairment before and after surgery
Change of Mini-Mental State (MMS) test score | Change of MMS score between two time points (the day before surgery and 3h postoperatively
  Change of 30-point questionnaire that is used to measure cognitive impairment before and after surgery
Change of Mini-Mental State (MMS) test score | Change of MMS score between two time points (the day before surgery and 24h postoperatively
  Change of 30-point questionnaire that is used to measure cognitive impairment before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xia Shen, M.D., Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evered L, Scott DA, Silbert B, Maruff P. Postoperative cognitive dysfunction is independent of type of surgery and anesthetic. Anesth Analg. 2011 May;112(5):1179-85. doi: 10.1213/ANE.0b013e318215217e. Epub 2011 Apr 7. PMID 21474666
- [Background] Larsen B, Seitz A, Larsen R. Recovery of cognitive function after remifentanil-propofol anesthesia: a comparison with desflurane and sevoflurane anesthesia. Anesth Analg. 2000 Jan;90(1):168-74. doi: 10.1097/00000539-200001000-00035. PMID 10624999
- [Background] Royse CF, Andrews DT, Newman SN, Stygall J, Williams Z, Pang J, Royse AG. The influence of propofol or desflurane on postoperative cognitive dysfunction in patients undergoing coronary artery bypass surgery. Anaesthesia. 2011 Jun;66(6):455-64. doi: 10.1111/j.1365-2044.2011.06704.x. Epub 2011 Apr 18. PMID 21501129
- [Background] Roy S, Smith LP. Surgical fires in laser laryngeal surgery: are we safe enough? Otolaryngol Head Neck Surg. 2015 Jan;152(1):67-72. doi: 10.1177/0194599814555853. Epub 2014 Oct 24. PMID 25344591